CLINICAL TRIAL: NCT02522546
Title: A Study to Assess the Carriage of Pneumococci in Children Aged 1-5 Years, and Their Household Contacts
Acronym: PIN
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Principal Investigator, Prof. Elizabeth Miller, Prof Elizabeth Miller, Public Health England
Other Study IDs: PIN
Record Dates: First submitted 2015-07-22; First posted 2015-08-13 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-08

CONDITIONS: Nasal Carriage of Pneumococci

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- nasopharyngeal swab: Children ages 1-5 years and their household contacts
  Interventions: Other: nasopharyngeal swab

INTERVENTIONS:
Other: nasopharyngeal swab — nasopharyngeal swab
  Other Names: nose swab

SUMMARY:
Pneumococci are bacteria which can cause serious and potentially life threatening illnesses like meningitis and blood poisoning.

Pneumococcal vaccines (PCV) have been given in the national immunisation schedule since 2006.Carriage studies allow assessment of how the strains in the nose change over time, in that by clearing some strains away which other strains take up those niches in their place both in children and in their close/household contacts. This helps to inform the best use of the vaccines available and for future vaccine development and which strains would be useful to include.

DETAILED DESCRIPTION:
Pneumococci are bacteria which can cause serious and potentially life threatening illnesses like meningitis and blood poisoning. There are ~90 strains, some are more dangerous than others in the severity of the disease they cause. Around half of all children carry pneumococci at the back of their nose without any ill effect. Pneumococcal vaccines (PCV) have been given in the national immunisation schedule since 2006. Vaccines protect individuals by making antibodies to be made in the blood and these vaccines help to clear the pneumococci from the nose, which helps control disease in the population by stopping their onward transmission when children cough and sneeze. This clearing effect is specific to the strains that are included in the vaccine. The first vaccines used included seven (PCV7) strains and the one used currently includes 13 (PCV13).

This group has conducted three previous carriage studies, and this will be the fourth. The first was before any vaccine was used, the second just after PCV7 was introduced and the third after the UK moved to using PCV13. These carriage studies allow assessment of how the strains in the nose change over time, in that by clearing some strains away which other strains take up those niches in their place both in children and in their close/household contacts. This helps to inform the best use of the vaccines available and for future vaccine development and which strains would be useful to include.

All families registered at participating surgeries, with a child aged 1-5 years, will be invited to take part. The study involves a single nasopharyngeal swab and a saliva swab from the child and as many other household members as are happy to participate. Participants may be seen at their GP surgery or in the home if more mutually convenient

ELIGIBILITY:
Inclusion Criteria:

* At least one child aged 1 to 5 years in the household
* Written informed consent obtained from the child's parent / legal guardian for their participation, and for any participating household contacts

Exclusion Criteria:

* Moderate to severe cerebral palsy or other debilitating condition
* Syndromes and neurological disorders affecting swallowing.
* Ear, nose & throat disorders affecting local anatomy for swabbing (e.g. malformed ears)
* Confirmed or suspected immunodeficiency (congenital or acquired) or receiving immunosuppressive therapy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children aged 1-5 years and their household contacts
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
pneumococcal carriage rate in children aged 1-5 years, older children and adolescents (aged 5-20 years) and adults (aged >20 years), five years after the introduction of PCV13 | baseline
  pneumococcal carriage rates for PCV13 and non-PCV13 serotypes in children aged 1-5 years, older children and adolescents (aged 5-20 years) and adults (aged >20 years), five years after the introduction of PCV13.
invasiveness of any emerging replacement carriage serotype | baseline
  invasiveness of any emerging replacement carriage serotypes by estimating case: carrier ratio (CCR) using national surveillance data for invasive pneumococcal disease

SECONDARY OUTCOMES:
carriage rates of individual serotype | baseline
changes in carriage serotype | baseline
  changes in carriage serotype, by age, vs previous carriage studies performed by the Health Protection Agency in 2001/02, 2008/09 and 2012 in children and adults. This includes changes in the prevalence of proportion and changes in the proportion of carriage strains that are vaccine and non-vaccine types

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD — Public Health England
Locations (2):
- United Kingdom (2):
  - Gloucestershire primary care, Gloucestershire, Gloucestershire
  - Hertfordshire primary care, Hertfordshire, Hertfordshire

REFERENCES:
- [Result] Southern J, Andrews N, Sandu P, Sheppard CL, Waight PA, Fry NK, Van Hoek AJ, Miller E. Pneumococcal carriage in children and their household contacts six years after introduction of the 13-valent pneumococcal conjugate vaccine in England. PLoS One. 2018 May 25;13(5):e0195799. doi: 10.1371/journal.pone.0195799. eCollection 2018. PMID 29799839
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/29799839